CLINICAL TRIAL: NCT01508416
Title: Study of Thrombin Generation During the 3 First Cycles of Chemotherapy in Patients With Newly Diagnosed Multiple Myeloma: a Multicentric Study
Brief Title: Study of Thrombin Generation During the 3 First Cycles of Chemotherapy in Patients With Newly Diagnosed Multiple Myeloma
Acronym: METRO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other); Groupe de Recherche sur la Thrombose (Other)
Responsible Party: Sponsor
Other Study IDs: 1108178; 2011- A01529-32 (Other: Afssaps)
Record Dates: First submitted 2011-12-15; First posted 2012-01-12 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Newly diagnosed; Thrombin generation; TFPI; Tissue Factor pathway inhibitor; Protein S; Thrombosis; Chemotherapy
MeSH Terms: conditions — Multiple Myeloma; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Multiple Myeloma: Patients with newly diagnosed Multiple Myeloma required chemotherapy

SUMMARY:
Patients with Multiple Myeloma (MM) are at increased risk of venous thromboembolic event, especially in newly diagnosed patients and during induction treatment with thalidomide in combination with dexamethasone. This association was mainly heightened during the 3 first months of chemotherapy.

Several coagulation abnormalities have been described. Laboratory tests measuring the overall thrombophilic tendency might be useful to assess thrombosis risk.

The aim of this study is to compare thrombin generation by calibrated automated thrombogram during the 3 first cycles of chemotherapy in patients with newly diagnosed MM.

ELIGIBILITY:
Inclusion Criteria:

* Inscription to medical assurance
* Patients who gave their written consent
* Patients with newly diagnosed Multiple Myeloma required chemotherapy

Exclusion Criteria:

* Patients with renal failure who need to undergo hemodialysis
* Patients with indication for curative anticoagulant therapy
* Patient with 3 month follow-up not possible
* Patient with life expectancy < 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed Multiple Myeloma required chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in Thrombin generation measure | day 21
  change from baseline in Thrombin generation measure
change from baseline in Thrombin generation measure | day 42
  change from baseline in Thrombin generation measure
change from baseline in Thrombin generation measure | day 63
  change from baseline in Thrombin generation measure
change from baseline in Thrombin generation measure | day 0
  change from baseline in Thrombin generation measure

SECONDARY OUTCOMES:
image-confirmed venous thromboembolic events | day 63
  Estimate the incidence of venous thromboembolic events until day 63
change from baseline in TFPI resistance measure | day 21
  change from baseline in TFPI resistance measure
change from baseline in acquired protein S deficiency measure | day 21
  change from baseline in acquired protein S deficiency measure
change from baseline in TFPI resistance measure | day 42
  change from baseline in TFPI resistance measure
change from baseline in TFPI resistance measure | day 63
  change from baseline in TFPI resistance measure
change from baseline in acquired protein S deficiency measure | day 42
  change from baseline in acquired protein S deficiency measure
change from baseline in acquired protein S deficiency measure | day 63
  change from baseline in acquired protein S deficiency measure
change from baseline in TFPI resistance measure | day 0
  change from baseline in TFPI resistance measure
change from baseline in acquired protein S deficiency measure | day 0
  change from baseline in acquired protein S deficiency measure

CONTACTS AND LOCATIONS:
Overall Officials: Bernard TARDY, MD-PhD, Principal Investigator — CHU de Saint-Etienne - CIC-EC (CIE3)
Locations (5):
- France (5):
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de Nancy, Nancy
  - Service de Médecine Interne - CHU de Saint Etienne, Saint-Etienne
  - Service de rhumatologie - CHU de Saint Etienne, Saint-Etienne
  - Service d'hématologie - ICL, Saint-Priest-en-Jarez